CLINICAL TRIAL: NCT05861466
Title: Comparative Study Between Intravitreal Injection of Ranibizumab with and Without Prior Anterior Chamber Paracentesis in Patients with Diabetic Macular Oedema Using Optical Coherence Tomography Angiography [OCT-A]
Brief Title: Comparative Study Between IVI of Ranibizumab with and Without Prior ACP in Patients with DME Using OCT-A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Sanad, Assistant lecturer of ophthalmology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD 1692022
Record Dates: First submitted 2023-05-02; First posted 2023-05-16 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Patients with eyes with non ischemic diffuse center involving DME will be assigned to receive IVI of ranibizumab without Anterior Chamber Paracentesis.
  Interventions: Drug: intra-vitreal injection of Ranibizumab
- Group B (Active Comparator): Patients with eyes with non ischemic diffuse center involving DME will be assigned to receive IVI of ranibizumab with Anterior Chamber Paracentesis.
  Interventions: Drug: intra-vitreal injection of Ranibizumab; Procedure: anterior chamber paracentesis

INTERVENTIONS:
Drug: intra-vitreal injection of Ranibizumab — The intravitreal injection will be performed with ranibizumab (0.5 mg/0.05 mL through a 27-gauge needle that will be inserted into the sclera 3.5 mm from the corneal limbus in pseudophakic patients, and 4 mm in phakic patients.
Procedure: anterior chamber paracentesis — A 27-gauge needle on a 1-mL syringe will be inserted into the anterior chamber of the eye, and approximately 0.05 mL of aqueous humor will be withdrawn.
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to to evaluate the changes in retinal microvasculature secondary to intra-ocular pressure changes post intra-vitreal injection in patients with diabetic macular oedema highlighting the effect of prior anterior chamber paracentesis on such changes if present .

The main question[s]it aims to answer are:

•[is there any effect of post intra-vitreal injection IOP spikes on retinal microvasculature?] •[is there any effect of Prior Anterior Chamber Paracentesis?] Participants in group A will be subjected to an identified approved treatment( intra-vitreal injection)& Participants in group B will be subjected to a prior ACP with the intra-vitreal injection . ]

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus type II.
* Patients with visual acuity > 0.1, able to fixate and with clear visual media.
* Patients with eyes with non ischemic diffuse center involving DME were randomly assigned to receive IVI of ranibizumab either without (group A) or with (group B) ACP.

Exclusion Criteria:

* Age under 40 years.
* Poorly controlled diabetics (HbA1C greater than 9.0%)
* Proliferative diabetic retinopathy.
* OCT-Angiographic evidence of ischemia (enlarged foveal avascular zone, paramacular areas of capillary nonperfusion)
* Neovascular AMD in the study eye.
* History of glaucoma.
* Tilted disc and optic disc anomalies.
* One-eyed patients.
* Usage of systemic or topical corticosteroids.
* Patients with a history of intraocular surgery other than cataract surgery.
* Systemc diseases rather than hypertension and diabetes mellitus.
* Corneal opacities that might hinder acquisition of good quality OCT images.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
the acute change in angiographic parameters | 1 day
  OCTA of macula and peripapillary region with documentation of vessel density

SECONDARY OUTCOMES:
the acute change in intra-ocular pressure | 1 day
  Goldman applanation tonometry for evaluation of IOP

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No